CLINICAL TRIAL: NCT01594424
Title: A Phase I/II Trial of Tocilizumab + Intravenous Immunoglobulin (IVIG) as Agents to Reduce Donor-Specific Anti-HLA Antibodies (DSA) and Improve Transplant Rates in Highly-HLA Sensitized Patients Awaiting Kidney Transplantation
Brief Title: A Safety Study of Tocilizumab to Improve Transplant Rates in Highly Sensitized Patients Awaiting Kidney Transplantation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Stanley Jordan, MD, Medical Director, Medical Director, Renal Transplantation & Transplant Immunotherpay, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Actemra + IVIG
Record Dates: First submitted 2012-05-04; First posted 2012-05-09 (Estimated); Results first posted 2015-08-05 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-07

CONDITIONS: End Stage Renal Disease (ESRD)
Keywords: Donor-Specific Anti-HLA Antibodies; Kidney Transplantation
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — tocilizumab; Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IVIG + Tocilizumab (Experimental)
  Interventions: Drug: Tocilizumab; Drug: Intravenous Immunoglobulin

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab 8mg/kg on Days 0, 15, 30, 45, 75, 105, 119, 135, 149, and 180
  Other Names: Actemra®
Drug: Intravenous Immunoglobulin — All HS who meet criteria for desensitization will receive IVIG 10% (2.0 g/kg [maximum 140 g per dose] on days 1 and 30).
  Other Names: IVIG

SUMMARY:
In this Phase I/II trial, 10 highly sensitized patients will be entered after informed consent and will receive Intravenous Immunoglobulin (IVIG) at 2 gm/kg + Tocilizumab 8 mg/kg x 5 doses on days 15, 45, 75, 105, 119, 135, and 149. If robust reductions in anti-HLA antibody are seen, patients will progress to kidney transplantation when an "acceptable" crossmatch is achieved with a living donor (LD) or deceased donor (DD). Those receiving transplants will also receive Tocilizumab infusion monthly X7 doses post-transplant. All subjects will have intensive monitoring of Donor Specific Antibodies (DSA), viral PCRs, and routine post-transplant labs. At 6 months post-transplant, those who have retained their transplanted kidney will have a protocol biopsy.

ELIGIBILITY:
Inclusion Criteria:

* End-stage renal disease.
* No known contraindications for therapy with IVIG 10%/Actemra®.
* Age 18-65 years at the time of screening.
* CPRA > 50% demonstrated on 3 consecutive samples, UNOS wait time sufficient to allow DD offers, history of sensitizing events, positive crossmatch with the intended donor. LDs with DSA and Crossmatch positivity.
* Subject/Parent/Guardian must be able to understand and provide informed consent.

Exclusion Criteria:

* Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months following randomization.
* Treatment with any investigational agent within 4 weeks (or 5 half-lives of the investigational drug, whichever is longer) of screening.
* Previous treatment with any cell-depleting therapies, including investigational agents or approved therapies, some examples are CAMPATH, anti-CD4, anti-CD5, anti¬CD3, anti-CD19 and anti-CD20 within 6 months of baseline.
* Treatment with intravenous gamma globulin, plasmapheresis or Prosorba column within 6 months of baseline
* Immunization with a live/attenuated vaccine within 2 months prior to baseline.
* Previous treatment with TCZ (an exception to this criterion may be granted for single dose exposure upon application to the sponsor on a case-by-case basis).
* Any previous treatment with alkylating agents such as chlorambucil, (within 1 year) or with total lymphoid irradiation.

Exclusions for General Safety:

* History of severe allergic or anaphylactic reactions to human, humanized or murine monoclonal antibodies.
* Evidence of serious uncontrolled concomitant cardiovascular, nervous system, pulmonary (including obstructive pulmonary disease), hepatic, endocrine (include uncontrolled diabetes mellitus) or gastrointestinal disease (including complicated diverticulitis, ulcerative colitis, or Crohn's disease.)
* Current liver disease as determined by principal investigator unless related to primary disease under investigation
* Known active current or history of recurrent bacterial, viral, fungal, mycobacterial or other infections (including but not limited to tuberculosis and atypical mycobacterial disease, Hepatitis B and C, and herpes zoster, but excluding fungal infections of nail beds). These are limited to non-access related infections.
* Any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks prior to screening.
* Active TB requiring treatment within the previous 3 years. Patients should be screened for latent TB and, if positive, treated following local practice guidelines prior to initiating TCZ. Patients treated for tuberculosis with no recurrence in 3 years are permitted.
* Primary or secondary immunodeficiency (history of or currently active) unless related to primary disease under investigation.
* Evidence of active malignant disease, malignancies diagnosed within the previous 10 years (including hematological malignancies and solid tumors, except basal and squamous cell carcinoma of the skin or carcinoma in situ of the cervix uteri that has been excised and cured), or breast cancer diagnosed within the previous 20 years unless related to primary disease under investigation.
* Pregnant women or nursing (breast feeding) mothers.
* Patients with reproductive potential not willing to use an effective method of contraception.
* History of alcohol, drug or chemical abuse within 1 year prior to screening.
* Neuropathies or other conditions that might interfere with pain evaluation unless related to primary disease under investigation.
* Patients with lack of peripheral venous access.
* Body weight of > 150 kg.

Laboratory Exclusion criteria (at screening):

* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 1.5 times upper limit of normal (ULN)
* Total Bilirubin > ULN
* Platelet count < 100 x 109/L (100,000/mm3)
* Hemoglobin < 85 g/L (8.5 g/dL; 5.3 mmol/L)
* White Blood Cells < 3.0 x 109/L (3000/mm3)
* Absolute Neutrophil Count < 2.0 x 109/L (2000/mm3)
* Absolute Lymphocyte Count < 0.5 x 109/L (500/mm3)
* Positive Hepatitis BsAg, or Hepatitis C antibody

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-06; Primary Completion 2014-11 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Jordan, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] Vo AA, Choi J, Kim I, Louie S, Cisneros K, Kahwaji J, Toyoda M, Ge S, Haas M, Puliyanda D, Reinsmoen N, Peng A, Villicana R, Jordan SC. A Phase I/II Trial of the Interleukin-6 Receptor-Specific Humanized Monoclonal (Tocilizumab) + Intravenous Immunoglobulin in Difficult to Desensitize Patients. Transplantation. 2015 Nov;99(11):2356-63. doi: 10.1097/TP.0000000000000741. PMID 26018350

RESULTS

PARTICIPANT FLOW:
Groups:
- IVIG + Tocilizumab (TCZ): All patients received IVIg 10% (2.0 g/kg [maximum 140 g per dose] on days 1 and 30) and TCZ (8 mg/kg administered on day 15, then monthly for 6 months). If transplanted, patients received IVIg on day 0; TCZ on day 2 and TCZ monthly for 6 months patients received alemtuzumab 30 mg subcutaneously x1 dose as induction and were maintained on triple regimen with tacrolimus (target level of 7 to 9 ng/mL in first 6 months; then 5-7 ng/mL between 6 and 12 months; then 3-5 ng/mL thereafter); mycophenolate mofetil and prednisone taper.
Period: Overall Study
Arm/Group | IVIG + Tocilizumab (TCZ)
Started | 10
Completed | 8
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | IVIG + Tocilizumab (TCZ)
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Infectious Complications Following Transplantation
Description: patients will be in the study for up to 2 years
Time Frame: 24 months
Measure: Number; unit: participants
Arm/Group | IVIG + Tocilizumab (TCZ)
Number analyzed (Participants) | 10
participants | 2

ADVERSE EVENTS:
Groups:
- IVIG + Tocilizumab: All patients received IVIg 10% (2.0 g/kg [maximum 140 g per dose] on days 1 and 30) and TCZ (8 mg/kg administered on day 15, then monthly for 6 months). If transplanted, patients received IVIg on day 0; TCZ on day 2 and TCZ monthly for 6 months patients received alemtuzumab 30 mg subcutaneously x1 dose as induction and were maintained on triple regimen with tacrolimus (target level of 7 to 9 ng/mL in first 6 months; then 5-7 ng/mL between 6 and 12 months; then 3-5 ng/mL thereafter); mycophenolate mofetil and prednisone taper.
Arm/Group | IVIG + Tocilizumab
Serious Adverse Events (participants affected / at risk) | 4/10
Other Adverse Events (participants affected / at risk) | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IVIG + Tocilizumab (N=10)
Pneumonia (Infections and infestations) | 1 (1) — Fluid overload and pulmonary congestion as a result of underdialysis
Hyperkalemia (Renal and urinary disorders) | 1 (1) — Hyperkalemia in the same patient who had pneumonia
Infective colitis with colonic perforation (Gastrointestinal disorders) | 1 (1) — 1 transplanted patient developed infective colitis with colonic perforation required bowel resection (possibly related to study drug)
Bells Palsy (Infections and infestations) | 1 (1) — 1 transplanted patient
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IVIG + Tocilizumab (N=10)
Nausea (Gastrointestinal disorders) | 1 (1)
abdominal pain (Musculoskeletal and connective tissue disorders) | 1 (1) — During hemodialysis pre-transplant, with normal amylase and lipse
Headache (General disorders) | 1 (1)
Itching (Musculoskeletal and connective tissue disorders) | 1 (1)
Blurred Vision (Eye disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
elevated liver function enzymes (Hepatobiliary disorders) | 3 (3)
Elevated blood pressure (Cardiac disorders) | 1 (1)
Minimal infusion related reaction (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No